CLINICAL TRIAL: NCT01210443
Title: A Phase 3, Multi-Center, Open Label Study To Evaluate The Long-Term Safety Of Sitaxentan Sodium In Japanese Subjects With Pulmonary Arterial Hypertension
Brief Title: Long-Term Open-Label, Safety Study Of Sitaxentan Sodium In Japanese Pulmonary Arterial Hypertension Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1321053
Record Dates: First submitted 2010-08-11; First posted 2010-09-28 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension, Pulmonary
Keywords: sitaxentan sodium pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — sitaxsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sitaxentan treatment (Experimental)
  Interventions: Drug: Sitaxentan

INTERVENTIONS:
Drug: Sitaxentan — sitaxentan sodium 100 mg

SUMMARY:
The safety and efficacy at 100 mg once daily for oral dose of sitaxentan sodium were demonstrated in the STRIDE clinical trial program. Sitaxentan sodium was approved in the EU, Canada and Australia. In this study, the long-term safety and efficacy after administrations of sitaxentan sodium at a dose of 100 mg alone or in combination with another medication will be investigated in Japanese PAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject who completed the B1321052 study as planned.

Exclusion Criteria:

* Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure >160 mm Hg or sitting diastolic blood pressure >100 mm Hg at Screening.
* Has hypotension defined as systolic arterial pressure <90 mm Hg after sitting for 5 minutes at Screening.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321053&StudyName=Long-Term%20Open-Label%2C%20Safety%20Study%20Of%20Sitaxentan%20Sodium%20In%20Japanese%20Pulmonary%20Arterial%20Hypertension%20Patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received one 100 mg film-coated tablet of sitaxentan daily for 12 weeks in preceding B1321052 study.
Groups:
- Sitaxentan Treatment: All participants received one 100 mg film-coated tablet of sitaxentan daily. The intended treatment period was until sitaxentan was launched in Japan. Participants could receive additional PAH-specific drug treatment (beraprost or sildenafil) at the discretion of the investigator.
Period: Overall Study
Arm/Group | Sitaxentan Treatment
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study terminated by sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 2
Age, Customized [Number; unit: Participants]
  <=18 years | 0
  19-64 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, severe adverse events, serious adverse events
Time Frame: Up to 22 days (last participant discontinuation)
Population: The safety analysis set is defined as all subjects who receive at least one dose of study drug during this extension study.
Measure: Number; unit: Participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 2
Participants
  Treatment emergent all-causality adverse events | 1
  Treatment emergen-causality serious adverse events | 0
  Treatment emergent all-causality severe adverse ev | 0

2. Secondary Outcome: Percentage of Participants With Clinical Worsening
Description: Clinical worsening is defined as 1) Hospitalization for worsening pulmonary arterial hypertension, 2) On-study death, 3) Heart-lung or lung transplantation, 4) Atrial septostomy, 5) Addition of the chronic medications for the treatment of worsening pulmonary arterial hypertension, and 6) Initiation of oxygen.
Time Frame: Up to 22 days (last participant discontinuation)
Population: The efficacy analysis set was defined as all subjects who receive at least one dose of study drug during this extension study and have efficacy observations at baseline of the preceding study (B1321052) in any efficacy assessments.
  Descriptive statistics for any efficacy endpoints were not calculated due to a small number of participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance
Description: Change from baseline in 6-minute walk distance is calculated as the value at each time point (every 12 weeks until Week 48 and every 24 weeks after Week 48) minus value at baseline.
Time Frame: Up to 22 days (last participant discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Change From Baseline in WHO Functional Class
Description: The change from baseline in WHO functional class was classified into "Improved", "No change" and "Worsened". The change from baseline in WHO functional class is summarised with percentage of participants at each time point (every 12 weeks until Week 48 and every 24 weeks after Week 48).
Time Frame: Up to 22 days (last participant discontinuation)
Population: as for outcome 2
Measure: Number; unit: Parcentage of participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Blood Concentration of N-amino Terminal Fragment of the Prohormone Brain Natriuretic Peptide (NT-pro BNP)
Description: Change from baseline in Blood Concentration of NT-pro BNP is calculated as the value at each time point (every 12 weeks until Week 48 and every 24 weeks after Week 48) minus value at baseline.
Time Frame: Up to 22 days (last participant discontinuation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxentan Treatment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxentan Treatment (N=2)
Diarrhoea (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.